CLINICAL TRIAL: NCT07085377
Title: Autonomous Methadone Delivery System by Nurses
Acronym: DIADEME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL23_0905
Record Dates: First submitted 2025-06-26; First posted 2025-07-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder (OUD); Addictology
Keywords: Opioid use disorder (OUD); Methadone; Autonomous nursing system medication delivery; Nursing Care Delivery System
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: A multicenter prospective open-label randomized (patient), controlled superiority trial, in two parallel-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient DIADEME group (Experimental): The patient DIADEME group corresponds to the autonomous nursing system for managing the dispensing of methadone. This standardized protocol, in line with best practice guidelines, enables doses to be adjusted by nurses on the basis of a clinical assessment scheme incorporating the state of opioid withdrawal and overdosing.
  Interventions: Procedure: DIADEME strategy; Procedure: Individual semi directive interview
- Patient control group (Other): The patient control group is managed in accordance with standard practice guidelines for patients with OUD, with care pathway provided by the hospital practictioner, assisted by nursing team.
  Interventions: Procedure: Controle strategy
- Healthcare professionals group (Other): Focus groups with healthcare professionals will be held in each CSAPA after the last patient has been included in the center.
  Each focus group will consist of 6 to 8 professionals, including nurses and doctors involved in implementing the care protocol
  Interventions: Procedure: Individual semi directive interview

INTERVENTIONS:
Procedure: DIADEME strategy — This strategy consists of implementing the standardized DIADEME protocol. It, in line with best practice recommendations, enables nurses to adjust methadone dosage on the basis of a clinical assessment scheme incorporating opioid withdrawal and overdosing and includes:
  * initial medical consultation with the hospital practitioner for an addictology and psychiatry assessment, OUD assessment, and initial prescription of methadone for 3 months
  * ECG prior to any methadone prescription, hepatitis B, C, HIV testing may be offered, and an emergency NALOXONE kit will be given to the patient or prescribed
  * follow-up consultations with an nurse at least every 7 days, and more frequently if necessary.Dosages can be adjusted by the nurse on the basis of the standardized DIADEME protocol
  * medical consultation are only in the event of major withdrawal symptoms or overdosing or in the event of any incident not covered by the protocol and warranting rapid medical advice or at the patient's request
  Arms: Patient DIADEME group
Procedure: Controle strategy — The control strategy corresponds to standard practice guidelines for patients suffering from drug addiction, with the care pathway provided by the hospital practitioner, assisted by the nursing team.
  Arms: Patient control group
Procedure: Individual semi directive interview — Individual semi-directive interviews with a sample of patients from the DIADEME group (2 to 3 volunteer patients per CSAPA for a total of 20 to 30 interviews) will be conducted by a research psychologist and carried out at one month after the end of follow-up (3 months).
  Themes covered will include: commitment to care, patient/professional relationship, understanding of follow-up and treatment, experience of care and services at the addictology center, satisfaction with services received, level of response to expectations).
  Individual semi-directive interviews with a sample of healthcare professionals focus group will be also conducted by a research psychologist and carried out after the last patient has been included in the center. The aim will be to understand the effects of the intervention and identify its impact on professionals and the organization of the centers.
  Arms: Healthcare professionals group; Patient DIADEME group

SUMMARY:
Initiations of methadone treatment for opiode use disorder (OUD) are carried out in France in specialized centers, known as centers for care, support and prevention in addictology (CSAPA) In this way, hospital practitioners initiate the prescription of methadone, which is delivered on the spot by the nursing team. CSAPA nurses, and addictology nurses more generally, have a real range of skills which can include adapting treatment doses according to a protocol pre-established in a team, and medically validated (French law no. 2019-774 of July 24, 2019 relating to the organization and transformation of the healthcare system).

The methadone speciality used for initiation in CSAPAs is almost always the syrup form. The capsule form can only be used after one year's treatment, unless exceptionally authorized by the medical officer of the French National Health Insurance Fund. However, regulations stipulate that the prescription of methadone syrup must be renewed every fourteen days, which in theory means that a CSAPA doctor must see the patient at least twice a month to renew the prescription, throughout the entire course of treatment.

In practice, medical resources are often not sufficient for patients to be seen by a doctor at such a rate. Numerous palliative organizations exist, though they remain poorly described and documented. In some centers, doctors focus primarily on initiations, and prescriptions for patients for whom "stability" has been achieved are sometimes renewed for longer periods than fourteen days, with nurses in charge of assessing whether this organization is suitable for the patient. The notion of stability varies significantly from one center to another, and may mean achieving a constant dose, stopping illicit opioid use, or other criteria more focused on the patient's psychosocial reintegration. By outlining the missions of Addictology nurses, and more specifically of CSAPA nurses, the investigators can define the essential skills required of nurses to carry out these missions.

The main hypothesis of the DIADEME study is that semi-autonomous management of methadone treatment initiation by CSAPA nursing teams helps to reinforce adherence to care and thus improve retention rates in the 3 months following initiation.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years of age or older,
* With opioid use disorder (OUD) according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria (other authorized psychoactive substance use),
* Intending to start methadone treatment for OUD in a CSAPA center within 7 days,
* Agreeing to be followed up in a CSAPA over the next 3 months,

Exclusion Criteria:

* Having taken methadone treatment (on prescription) in the three months prior to inclusion,
* Simultaneous medical care in another addictology facility,
* with a day-hospital project,
* Referral to town prescriber or town pharmacy planned and/or requested by patient before 3 month,
* Non-stabilized psychiatric disorder or cognitive impairment likely to compromise compliance and involvement in care (at investigator's discretion),
* Inability to communicate and express themselves in French language,
* Subject to a legal protection measure other than curatorship,
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-04-08 (Estimated); Study Completion 2028-04-08 (Estimated)

PRIMARY OUTCOMES:
Patient retention in care | 3 months
  Patient retention in care at 3 months, defined as the last two methadone dispensing appointments honored in the 15 days preceding the end of the study (3 months), in the absence of a documented situation that prevented the patient from honoring his appointments (death, hospitalization, etc.).

SECONDARY OUTCOMES:
Euroqol EQ-5D 5 (EuroQol-5 Dimensions, 5 Levels Questionnaire) score | 3 months
  The outcome criterion for cost-utility analysis is the number of quality-adjusted life years (QALYs) gained. QALYs will be estimated on the basis of responses to the Euroqol EQ-5D 5L scale.
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the 5 dimensions.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
  The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Medical cost of each strategy (DIADEME and Controle strategy) | 3 months
  Budgetary impact for funders of extending the system to all CSAPAs in France (if efficiency is demonstrated).
  Costs of medical and nursing consultations, care for adverse events, i.e. consultations and hospitalizations, particularly in connection with OST misuse.
Opioid withdrawal | At 2 and 3 months
  Opioid withdrawal is described as the declared absence of opioid use (excluding methadone) with negative urinary toxins (excluding methadone and degradation products)
CSQ-8 (Client Satisfaction Questionnaire) score | 3 months
  Patients' overall satisfaction with CSAPA is assesed using the CSQ-8 scale (Client Satisfaction Questionnaire) The CSQ-8 scale consists of 8 questions that assess aspects like quality of service, whether patients' needs were met, likelihood of recommending the program, and overall satisfaction. Patients are asked to rate statements on a 4-point scale and are invited to provide additional comments.
Total methadone doses | over the 3-month follow-up period
  Total methadone doses delivered and related to follow-up time (mg er day) during the follow-up period
Overdose episode | At 1, 2 and 3 months
  Proportion of occurrences of at least one overdose episode (assessed clinically and by monthly patient declaration)
Hospital admissions | At 1, 2 and 3 months
  Proportion of all-cause hospital admissions (assessed on the basis of monthly patient declarations, or external data such as medical correspondence)
Adverse event | At 1, 2 and 3 months
  Proportion of occurrence and number of adverse events and serious adverse events (reported and assessed at each clinical evaluation point)
Opiate withdrawal | At 1, 2 and 3 months
  Proportion of patients with at least one moderate (>25) to severe (>36) opiate withdrawal assessed by the Clinical Opioid Withdrawal Scale (COWS)
Montgomery and Asberg Depression Rating Scale (MADRS) score | Between inclusion and 3 months
  Changes in severity of depression is assessed using the Montgomery and Asberg Depression Rating Scale score (MADRS) The Montgomery-Asberg Depression Rating Scale (MADRS) is a widely recognized clinical assessment tool designed to measure the severity of depressive episodes in patients with mood disorders.
  The scale consists of ten items, each targeting a different aspect of depression such as apparent sadness, reported sadness, inner tension, sleep disturbances, appetite, concentration, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored on a scale from 0 to 6, with higher scores indicating more severe symptoms. This scoring system allows clinicians to quantify symptoms in a standardized manner, facilitating both the initial assessment of depression severity and the ongoing monitoring of therapeutic interventions.
State-Trait Anxiety Inventory (STAI) score | Between inclusion and 3 months
  Changes in anxiety levels is assessed using the State-Trait Anxiety Inventory (STAI) scale.
  The State-Trait Anxiety Inventory (STAI) is a 40-item self-report measure of anxiety using a 4-point Likert-type scale (from 0 to 3 points) for each item. It has two scales: State anxiety, i.e. how one feels at the moment; and Trait anxiety, i.e. how one generally feels. Both scales consist of 20 items. The state scale has 10 reverse-scored items, the trait scale has 7.
Cannabis Use Disorder Identification Test - Revised (CUDIT-R) score | Between inclusion and at 1, 2 and 3 months
  Changes in cannabis use and use disorder is assesed using the Cannabis Use Disorder Identification Test - Revised (CUDIT-R) score. This questionnaire was designed for self-administration and is scored by adding each of the 8 items. Questions 1-7 are scored on a 0-4 scale. Question 8 is scored 0, 2 or 4.
Alcohol Use Disorders Identification Test (AUDIT-C) | Between inclusion and at 1, 2 and 3 months
  Assess changes in alcohol dependence using the Alcohol Use Disorders Identification Test (AUDIT-C).
Nicotine Dependence Test (FAGERSTROM) score | Between inclusion and at 1, 2 and 3 months
  Changes in nicotine consumption is assessed using the Nicotine Dependence Test (FAGERSTROM) scale.
  The Fagerstrom Nicotine Dependence Test is designed to provide an ordinal measure of nicotine dependence related to smoking. It contains six items that assess quantity of cigarettes smoked, compulsion to smoke and dependence. It is useful for screening for nicotine dependence and for assessing severity, which can be used for treatment planning and prognostic judgments.The lower is the score, the lower is the level of dependence.
Use of psychostimulant | Between inclusion and at 1, 2 and 3 months
  Assess the change in the proportion of psychostimulant use accurrence on patient declaration every month (if yes, type and frequency); Frequency will be measured by the following categories: daily consumption, several times/week, once/week, several times/month, 1 time/month
Fidelity of the DIADEME intervention | Up to 3 months
  Quantitative indicators describing compliance with the protocol implemented in CSAPAs (compliance with DIADEME protocol, number of nursing visits, delays, treatment adaptations carried out, requests for medical advice)
Acceptability of the DIADEME intervention | Up to 3 months
  Acceptability on the part of patients and professionals at participating centers, perceived effects of monitoring and adaptation of treatment by nursing staff, impact on patient care, professionals' perceptions of the new nursing role, obstacles and levers identified to sustain the intervention.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CSAPA, Association Bizia, Centre Hospitalier de la Côte Basque, Bayonne
  - CSAPA, Service d'Addictologie, Centre Hospitalier Charles Perrens, CHU de Bordeaux, Bordeaux
  - CSAPA de Brioude, Brioude
  - CSAPA, Association Nationale de Prévention en Alcoologie et Addictologie (ANPAA), Résidence Le Victor Hugo, Le Puy-en-Velay
  - CSAPA, Service Universitaire d'Addictologie de Lyon, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - CSAPA, Hôpital de la Croix Rousse, Hospices Civils de Lyon, Lyon
  - CSAPA, Service de Psychiatrie et d'Addictologie, Hôpital Civil, CHRU de Strasbourg, Strasbourg
  - CSAPA du Griffon, Oppelia Aria 69, Villeurbanne

IPD SHARING:
Plan to Share IPD: Undecided